CLINICAL TRIAL: NCT01736033
Title: A Multicenter, Randomized, Double-blind, Clinical Study to Investigate the Efficacy and Safety of Treatment With Tamsulosin 0.2mg Mono and Tamsulosin 0.2mg, Finasteride 5mg Combination Therapy in Patients With LUTS/BPH
Brief Title: Advanced Benefits of Alpha-blocker Monotherapy on Lower Urinary Tracts Symptoms(LUTS) Patients
Acronym: ABSOLUTE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry); Medical Research Collaborating Center, Seoul, Korea (Other)
Responsible Party: Principal Investigator, Soo Woong Kim, MD, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS1011
Record Dates: First submitted 2012-11-18; First posted 2012-11-29 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Benign Prostate Hyperplasia
Keywords: Lower Urinary Tracts Symptoms; 5 alpha reductase inhibitor; Proscar; Finasteride; alpha blocker; Tamsulosin; Harnal D
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin; Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamsulosin + Placebo (Placebo Comparator): Tamsulosin 0.2mg + Placebo 5 mg daily until clinical progression
  Interventions: Drug: Tamsulosin; Drug: Placebo
- Tamsulosin + Finasteride (Active Comparator): Tamsulosin 0.2mg + Finasteride 5 mg daily until clinical progression
  Interventions: Drug: Tamsulosin; Drug: Finasteride

INTERVENTIONS:
Drug: Tamsulosin — 1 tablet(0.2mg) orally q.d.
  Other Names: Harnal D (brand name in Asia); Flomax
Drug: Finasteride — 1 tablet(5mg) orally q.d.
  Other Names: Proscar
  Arms: Tamsulosin + Finasteride
Drug: Placebo — 1 tablet(0.2mg) orally q.d.
  Arms: Tamsulosin + Placebo

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of alpha-blocker monotherapy and alpha-blocker + 5-alpha reductase inhibitor combination therapy in benign prostate hyperplasia patients, and suggest guidelines of the combination therapy.

DETAILED DESCRIPTION:
Even though it should be decided on patients cautiously under careful consideration about prostate volume, Prostate Specific Antigen(PSA) level, symptom score and maximum uroflow, recently the combination therapy of alpha-blocker and 5-alpha reductase inhibitor has been tried imprudently in Korea.

As a result of several clinical trials which had conducted overseas for releasing the combination drug of alpha-blocker and 5-alpha reductase inhibitor, the superiority of the combination therapy has been proved, however, plenty of patients still don't derive additional profit from it.

Therefore, in this study, the investigators anticipate to meet with meaningful results on the clinical efficacy of alpha-blocker monotherapy and alpha-blocker + 5-alpha reductase inhibitor combination therapy in Korean benign prostate hyperplasia patients, and provide guidelines of the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged over 50
* Clinically diagnosed benign prostate hyperplasia(BPH)
* 8 ≤ IPSS ≤ 30
* 4 ml/sec ≤ Q max ≤ 15 ml/sec
* minimum voided volume ≥ 125 ml
* Post voided residual volume ≤ 250
* Volunteer who singed on informed consent documents

Exclusion Criteria:

* Past history of surgical procedure experience related to BPH
* Past history of taking 5-alpha reductase inhibitor(5-ARI) within 6 months before screening, or for more than 12 months regardless of the point of time
* Past history of taking alpha blocker within 2 weeks before screening
* Past history of acute urinary retention within 3 months before screening
* Serum PSA ≥ 10 ng/ml (but, in the case of 4 ng/ml ≤ PSA < 10 ng/ml, the patients can be included only if prostate cancer is excluded by prostate biopsy)
* Anatomical abnormalities of lower urinary tracts(urethrostenosis, diverticulosis, bladder neck contracture)
* Clinical status that affects voiding other than BPH(neurogenic bladder, Chronic Prostatitis/Chronic Pelvic Pain Syndrome, urinary infection, etc.)
* Unstable and significant medical condition including below

  * Unstable angina pectoris, myocardial infarction, cerebrovascular disease within 6 months before screening
  * Past history of malignant tumor including skin basal cell carcinoma within 5 years before screening
  * Medically uncontrollable diabetes mellitus, peptic ulcer disease
  * Severe hepatic diseases
  * Past history of renal failure or renal disease (serum creatinine > 1.4mg/dl)
  * Condition expected serious adverse event due to the investigational drug
* Other conditions considered not eligible for the trial upon investigator's judgement

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2012-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Progression | 1 & 2 months after baseline, and then every 3 months up to 4 years
  One of below
  * Deterioration of the symptoms
  * Acute urinary retention
  * Renal failure
  * Recurrent urinary tract infection
  * Urinary incontinence
  * Surgical procedure related to benign prostate hyperplasia

SECONDARY OUTCOMES:
International Prostate Symptom Score(IPSS) | 1 & 2 months after baseline, and then every 3 months up to 4 years
International Consultation on Incontinence Modular Questionnaire(ICIQ) male LUTS-short form | every 6 months up to 4 years
Uroflowmetry | every 6 months up to 4 years
  including Qmax, voided volume and post-void residual volume(PVR)
Prostate volume | every 1 year up to 4 years
Global Response Assessment(GRA) | every 1 year up to 4 years
PSA level | every 1 year up to 4 years
  PSA level will be examined in the central laboratory and be reported to each center as an adjusted number. It is because PSA level tends to decrease to 50% of baseline after taking finasteride for 1~4 years, so there is possibilities that the blindedness is broken with the actual result.
Blood Chemistry | every 1 year up to 4 years
  including Sodium, Potassium, Glucose, Urea nitrogen, Creatinine, ASpartate Transaminase(AST), ALanine Transaminase(ALT), Total bilirubin
Adverse Events | every visit up to 4 years
Physical examination | every 1 year up to 4 years
  Digital Rectal Exam, Breast exam
Male Sexual Health Questionnaire | every 6 months up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Soo Woong Kim, M.D., Principal Investigator — Seoul National University Hospital
Locations (11):
- South Korea (11):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheongnam-do
  - Hallym University Sacred Heart Hospital, Anyang, Gyeoggi
  - Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Eulji General Hospital, Seoul

REFERENCES:
- [Background] Shapiro E, Lepor H. Pathophysiology of clinical benign prostatic hyperplasia. Urol Clin North Am. 1995 May;22(2):285-90. PMID 7539174
- [Background] Garraway WM, Collins GN, Lee RJ. High prevalence of benign prostatic hypertrophy in the community. Lancet. 1991 Aug 24;338(8765):469-71. doi: 10.1016/0140-6736(91)90543-x. PMID 1714529
- [Background] Bosch JL, Kranse R, van Mastrigt R, Schroder FH. Reasons for the weak correlation between prostate volume and urethral resistance parameters in patients with prostatism. J Urol. 1995 Mar;153(3 Pt 1):689-93. doi: 10.1097/00005392-199503000-00039. PMID 7532234
- [Background] Chung TG, Chung J, Lee MS, Ahn H. Prevalence of benign prostatic hyperplasia in Jeong-Eup Area: community-based study. Korean J Urol 1999;40:52-8.
- [Background] The prevalence of benign prostatic hyperplasia in elderly men in Korea: a community-based study. Park HK, Park H, Cho S, Bae J, Jeong S, Hong SK, et al. Korean J Urol 2009;50:843-7.
- [Background] Lepor H, Gup DI, Baumann M, Shapiro E. Laboratory assessment of terazosin and alpha-1 blockade in prostatic hyperplasia. Urology. 1988 Dec;32(6 Suppl):21-6. PMID 2462301
- [Background] Noble AJ, Chess-Williams R, Couldwell C, Furukawa K, Uchyiuma T, Korstanje C, Chapple CR. The effects of tamsulosin, a high affinity antagonist at functional alpha 1A- and alpha 1D-adrenoceptor subtypes. Br J Pharmacol. 1997 Jan;120(2):231-8. doi: 10.1038/sj.bjp.0700907. PMID 9117115